CLINICAL TRIAL: NCT01602965
Title: Personalized Nutritional Program Plus a Nutritional Counseling Monthly Phone Call Versus a Personalized Nutritional Program With Self Help Informative Booklet
Brief Title: Effectiveness Between Nutritional Counseling Monthly Phone Call Versus Self Help Informative Booklet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0008363
Record Dates: First submitted 2012-05-04; First posted 2012-05-21 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Overweight
Keywords: obesity; counselling; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- counseling monthly phone calls (Experimental): the dietician will call the patient at home, and invite them to answer 11 open questions.The questionnaire collects information about weight loss, behaviours that need to be changed, problem-solving as to how to make the changes and physical activity levels.
  Interventions: Procedure: Counseling Monthly Phone Calls
- self help informative Booklet (Active Comparator): Self help informative booklet includes information on how to manage healthy weight, how to lose weight, physical activity and a simplified and abbreviated version of the main behavioural strategies.
  Interventions: Procedure: Self Help Informative Booklet

INTERVENTIONS:
Procedure: Counseling Monthly Phone Calls — the dietician will call the patient at home, and invite them to answer 11 open questions.The questionnaire collects information about weight loss, behaviors that need to be changed, problem-solving as to how to make the changes and physical activity levels.
  Arms: counseling monthly phone calls
Procedure: Self Help Informative Booklet — Self help informative booklet includes information on how to manage healthy weight, how to lose weight, physical activity and a simplified and abbreviated version of the main behavioural strategies
  Arms: self help informative Booklet

SUMMARY:
The purpose of this study is to evaluate the most effectiveness between a personalized nutritional program with a counseling monthly phone call Versus personalized nutritional program with self help Informative Booklet in a group of obesity or overweight patients without counseling phone call.

DETAILED DESCRIPTION:
Evaluate the best effectiveness between two methods applied in the Dietary Service of institute orthopedic Rizzoli for the achievement of the weight loss. Personalized nutritional program with counseling phone call versus personalized nutritional program with self help Informative Booklet in a controlled group.There will be compared two groups of patients: First group: patients subject to balanced personalized nutritional program associated to counseling monthly phone call ; compliance and loss of weight will be done monthly for one year. Second group: patients subject to balanced personalized nutritional program associated to self help informative Booklet; compliance and loss of weight will be done after six months and after one year from the first meeting.

ELIGIBILITY:
Inclusion Criteria:

* Female and male
* BMI >25 and <35
* Ages Eligible for Study: 18 years old to 75 years old
* Patients of the Institute Orthopedic Rizzoli subject to personalized nutritional program admitted to the wards and patients attending the clinic of Anaesthesiology, analgesic therapy, Rheumatology
* participants gave informed consent

Exclusion Criteria:

* Patients with psychiatric disorders (depression, bulimia, anorexia
* Concomitant use of medicines or food supplements that can alter the weight loss.
* Patients with inclusion criteria that have not signed the informative report and the declaration of consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Counseling Monthly Phone Calls | Self Help Informative Booklet
Started | 20 | 20
Completed | 16 | 18
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseling Monthly Phone Calls | Self Help Informative Booklet | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.08) | 56.5 (10.67) | 59.0 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 11 | 7 | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.94 (2.69) | 32.45 (2.41) | 32.69 (2.55)
Weight [Mean (Standard Deviation); unit: kg] | 96.15 (13.81) | 92.91 (9.95) | 94.53 (11.88)

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: The measure of weight must be detected with the help of a balance. Weight is measured using Professional Dial Column Scales without shoes or heavy clothing to the nearest 0.1 kg.
Time Frame: Percent Change in weight loss at one year
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | Counseling Monthly Phone Calls | Self Help Informative Booklet
Number analyzed (Participants) | 16 | 18
percentage of weight loss | 7.56 (5.42) | 2.80 (3.21)

ADVERSE EVENTS:
Arm/Group | Counseling Monthly Phone Calls | Self Help Informative Booklet
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No